CLINICAL TRIAL: NCT06451094
Title: Comparison of the Effectiveness of Ultrasound and Transfer Energy Capacitive and Resistive (TECAR) Therapy in Patients With Carpal Tunnel Syndrome
Brief Title: Effectiveness Transfer Energy Capacitive and Resistive Therapy in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-23-3833
Record Dates: First submitted 2024-06-03; First posted 2024-06-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Carpal Tunnel Syndrome; Energy Transfer Capacitative and Resistive Therapy
Keywords: Carpal tunnel syndrome; TECAR therapy; median nerve CSA
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US therapy, paraffin therapy (Experimental): Group 1, US therapy to the palmar region of the wrist, 5 minutes intermittently for 2 weeks, 5 times a week, for a total of 10 sessions and Paraffin therapy to the wrist area by dipping the hand 3 times into a paraffin bath and removing it, covering the entire wrist with paraffin, and waiting for 15 min (2 weeks, 5 times a week, for a total of 10 sessions).
  Interventions: Device: US therapy
- TECAR therapy, paraffin therapy (Experimental): Group 2, TECAR therapy to the palmar region of the wrist, 5 min capacitive (CAP) and 10 min resistive (RES), 3 days a week for 2 weeks, for a total of 6 sessions and Paraffin therapy to the wrist area by dipping the hand 3 times into a paraffin bath and removing it, covering the entire wrist with paraffin, and waiting for 15 min (2 weeks, 5 times a week, for a total of 10 sessions).
  Interventions: Device: TECAR

INTERVENTIONS:
Device: US therapy — 3 MHz probe with a BTL brand device at a dose of 1.5 watts/cm2 for 5 minutes intermittently for 2 weeks, 5 times a week, for a total of 10 sessions.
  Arms: US therapy, paraffin therapy
Device: TECAR — Transfer Energy Capacitative and Resistive Therapy
  Arms: TECAR therapy, paraffin therapy

SUMMARY:
Objective: The aim of this study was to evaluate the effect of Transfer Energy Capacitive and Resistive (TECAR) therapy on pain, symptom severity and function in patients diagnosed with carpal tunnel syndrome (CTS) based on clinical and electromyography (EMG) findings and to compare it with ultrasound therapy (US).

Methods: A total of 42 patients aged between 18 and 65 years, were randomly divided into two groups; group 1, US therapy 5 minutes intermittently for 2 weeks, 5 times a week, for a total of 10 sessions, group 2 TECAR therapy 5 min capacitive (CAP) and 10 min resistive (RES), 3 days a week for 2 weeks, for a total of 6 sessions. Both groups received paraffin therapy and wrist orthosis. All Patients were evaluated using the Visual Analog Scale (VAS) for pain and paresthesia levels, the Boston Carpal Tunnel Questionnaire (BCTQ) for symptom severity and functional levels. Additionally, median nerve CSA was measured by ultrasound, at the baseline, post-treatment, first and third months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over
* had pain and numbness in their hands for more than 3 months were evaluated
* Patients diagnosed with mild and moderate CTS by EMG

Exclusion Criteria:

* metabolic, rheumatic, or neurological diseases that could affect the median nerve cross-sectional area (CSA)
* patients who had previously undergone surgery on the wrist,
* oncology patients,
* pregnancy,
* pacemakers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | baseline (0 th day), after-treatment (15 th day), 1th month, 3rd month
  0 min , 10 is maximum pain score
Boston Carpal Tunnel Questionnaire (BCTQ) | baseline (0 th day), after-treatment (15 th day), 1th month, 3rd month
  symptom severity on functional tasks (Symptom Severity Scale), involving 11 items, and the other one on function status properly (Functional Status Scale), involving 8 items. Both subscales of BCTQ are scored between 1 and 5, and higher scores illustrate a greater degree of disability.

SECONDARY OUTCOMES:
Median nerve cross-sectional area (CSA) measurement | baseline (0 th day), after-treatment (15 th day), 1th month, 3rd month
  Median nerve CSA was measured by ultrasound on axial view at the scaphoid-pisiform level which is a reliable measurement for CTS. Three measurements were taken for analysis and the average value was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Özge TEZEN, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Tezen O, Ata AM, Uzun O, Cakir F, Yasar E. Comparison of the effectiveness of ultrasound and transfer energy capacitive and resistive (TECAR) therapy in patients with carpal tunnel syndrome. Lasers Med Sci. 2025 Mar 19;40(1):147. doi: 10.1007/s10103-025-04412-z. PMID 40106005